CLINICAL TRIAL: NCT06620029
Title: A Phase 1/2, Open-label Clinical Trial to Evaluate Safety and Efficacy of Combination Paclitaxel and BMX-001, in Adult Patients With Advanced, Recurrent, Metastatic Ovarian or Endometrial Cancer
Brief Title: BMX-001 + Paclitaxel in Adult Patients With Advanced, Recurrent, Metastatic Ovarian or Endometrial Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMimetix JV, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BMX-GyCa-001
Record Dates: First submitted 2024-09-18; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Ovarian Neoplasms; Endometrial Cancer, Endometrial Neoplasm
Keywords: BMX-001 plus Paclitaxel
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: Dose finding stage followed by an expansion cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMX-001 + PTX (Experimental): All patients will be administered BMX-001 + PTX weekly on Days 1, 8, 15, and 22 of each 28 day cycle. BMX-001 is a SC injection while PTX is IV.
  Interventions: Drug: BMX-001; Drug: Paclitaxel (Taxol)

INTERVENTIONS:
Drug: BMX-001 — BMX-001 consists of a porphyrin ring with pyridyl groups attached at each of the four methane bridge carbons. The nitrogen in the pyridyl ring is at the 2 position and has a side chain consisting of six carbons with an ether linkage. A manganese atom is chelated into the porphyrin ring and is the active center of the molecule. This molecule is an enzymatic scavenger of free radical species operating at close to diffusion-limited rates. BMX-001 (7-28 mg) will be given by subcutaneous (s.c.) injection starting on Day 1, Day 8, Day 15, and Day 22 of each 28-day PTX treatment cycle.
Drug: Paclitaxel (Taxol) — Paclitaxel will be given via IV infusion at a dose = 80 mg/m2 on Day 1, Day 8, Day 15, and Day 22 of each 28-day treatment cycle and will be sourced from standard commercial sources. Appropriate pretreatment prior to PTX will be given as per institutional standards. PTX management for any adverse event (AE) in any cycle, reasonably attributed to the chemotherapy agent that requires dose interruption should be managed per package insert, and/or institutional guidelines. Dose modification recommendations are provided in protocol to provide general consistency with dosing. Study Treatment dosing BMX-001 should continue even if the PTX is omitted. The subject may continue on PTX if the AE does not prohibit dosing per institutional practice. Grade 3 or higher infusion PTX reactions or recurrent infusion reactions may require permanent discontinuation of PTX. PTX may be continued in select patients using institutional desensitization protocol.

SUMMARY:
This research project addresses the urgent need for novel therapeutic strategies to overcome chemotherapy resistance and mitigate chemotherapy-induced peripheral neuropathy (CIPN) in patients with recurrent ovarian and endometrial cancers, which are among the most lethal gynecologic malignancies worldwide. The study focuses on BMX-001, a redox-active manganese metalloporphyrin compound that uniquely combines the ability to enhance anti-tumor efficacy and protect normal tissues from the toxic effects of chemotherapy, specifically paclitaxel (PTX). PTX, despite being a cornerstone of treatment, is associated with significant dose-limiting neurotoxicity, which severely impacts patients quality of life and limits the use of subsequent therapies. BMX-001 has demonstrated potential in preclinical models to not only augment the anti-tumor effects of PTX but also reduce PTX-induced neuropathy.

The research will be conducted through a single-site, Phase 1/2 clinical trial led by the Duke Cancer Institute. The trial aims to determine the recommended Phase 2 dose of BMX-001 when combined with weekly PTX and to evaluate the clinical activity of this combination therapy. Specifically, the trial will assess the safety, tolerability, and potential to double the dose of BMX-001, which is hypothesized to further enhance the efficacy of PTX without increasing toxicity. The study's specific aims include establishing the recommended dose for expansion, assessing objective response rates (ORR), and quantifying the reduction in PTX-induced neurotoxicity using validated questionnaires and monofilament testing. The project also incorporates the analysis of circulating tumor DNA (ctDNA) as a biomarker for treatment response, adding a layer of precision to the evaluation of the therapy response impact on tumor burden.

The outcomes of this research have the potential to significantly improve treatment protocols for patients with chemo-resistant gynecologic cancers by offering a therapy that enhances tumor control while protecting against debilitating side effects. Successful completion of this trial will lay the groundwork for larger, definitive trials and may extend the benefits of BMX-001 to other solid tumors, ultimately contributing to better survival outcomes and quality of life for a broader patient population.

DETAILED DESCRIPTION:
This clinical trial is a proof-of-concept Phase 1/2 study aimed at establishing the recommended Phase 2 dose (RP2D) of BMX-001 when administered in combination with weekly paclitaxel (PTX) in patients with advanced, metastatic ovarian or endometrial cancer. The rationale for this open-label trial is twofold: (1) response rates to weekly PTX in patients with platinum-resistant ovarian cancer (PROC) are generally low, and when a response is achieved, its duration is often short, necessitating novel therapeutic approaches to improve outcomes; (2) weekly PTX is associated with dose-limiting side effects, particularly chemotherapy-induced peripheral neuropathy (CIPN), which significantly impacts patients quality of life.

The trial includes a dose-finding stage designed to assess the safety and dose-limiting toxicities (DLTs) of the combination treatment. The study will use a Bayesian Optimal Interval (BOIN) design to test the safety of weekly BMX-001 injections in combination with weekly PTX. The goal is to determine if BMX-001 can be safely administered at increasing doses while enhancing both the efficacy of treatment as well as diminishing chemotherapy side effects in patients with recurrent, advanced ovarian and endometrial cancers.

Patients in the dose-escalation phase will receive up to 16 doses over an 8-week period. All participants will receive PTX at a dose of 80 mg/m² on the first day of each weekly cycle. The starting dose of BMX-001 will be 28 mg subcutaneously on the first day of each weekly cycle. Cohorts of three patients will be treated and evaluated for DLTs sequentially. If the starting dose is well-tolerated, subsequent cohorts will escalate to higher doses, with a maximum of 28 mg followed by 28 mg BMX-001 given 4-6 hours apart on the same day each week. Should any patients at Dose Level 1 experience DLTs, the dose will be de-escalated according to the BOIN design to Dose Level -1 (14 mg/week), and if necessary, further to Dose Level -2 (7 mg/week), which is the final de-escalation dose group.

Upon completion of the dose-finding phase, an expansion cohort will be enrolled at the RP2D. The study will enroll up to 27 patients in this trial. The primary outcome measure is to establish the RP2D of BMX-001 in combination with PTX. Secondary outcomes include evaluation of preliminary efficacy based on objective response rate (ORR) using RECIST v 1.1 per investigator assessment endpoints and obtaining a description of patient-reported outcomes of health related quality of life (HRQoL) quality of life (QoL) using FACT/GOG-NTX Questionnaire and monofilament testing.

Other outcome measures to be assessed in all patients include characterization of the pharmacokinetic profile of BMX-001 when delivered in combination with PTX in recurrent ovarian or endometrial cancer and also to assess correlations between B cell lymphoma/leukemia 2 (BCL2), Nrf2, TNF-alpha, and NFkB RNA and protein expression and activation, ctDNA, and clinical responses. This initial single arm trial is limited to 27 subjects based on the funds available in this SBIR. In spite of the small sample size, the study expects to obtain sufficient data to enable design a subsequent randomized trial that would meet registration requirements

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent advanced metastatic ovarian or endometrial cancer that progressed during or following prior SOC therapy
2. Aged 18 years or older
3. Eastern Cooperative Oncology Group performance status (ECOG-PS) of 0 to 1
4. Ability to understand and willingness to give written informed consent
5. Measurable disease according to RECIST v1.1 or assessable disease based on presence of malignancy pleural effusion or ascites, or disease that does not meet measurable criteria.
6. Negative serum pregnancy test within 48 hours of dosing if indicated.
7. Adequate bone marrow function
8. Adequate hepatic function
9. Adequate renal function as determined by calculated or measured creatinine clearance ≥30 mL/min (using Cockcroft- Gault equation) or serum creatinine < 1.5 X institutional ULN
10. Full recovery from all recent surgery on start date of treatment; at least 1 week must have elapsed from the time of a minor surgery (port placement at any time is acceptable); from the date of treatment at least 21 days must have elapsed from the time of a major surgery. Must have fully recovered from all surgery-related toxicities to Grade 1 or less
11. At least 28 days between termination of prior anticancer or hormonal therapy and first administration of BMX-001

Exclusion Criteria:

1. Residual Grade 2 peripheral neuropathy
2. Untreated central nervous system (CNS) metastases (surgery and/or radiotherapy), Subjects requiring corticosteroid therapy for the management of CNS metastases may not be on >10 mg/day prednisone or equivalent. Subjects that have demonstrated signs or symptoms of neurologic instability for 28 days or less prior to enrollment.
3. Is being treated with concurrent anticancer therapy or other interventional treatments administered for their underlying cancer
4. Subjects who have received prior therapy with weekly PTX in the recurrent setting.
5. Clinically significant cardiac disease.
6. History of or present CNS disease unrelated to cancer, unless adequately treated with standard medical therapy (eg, uncontrolled seizures)
7. Nonhealing wound, ulcer, or bone fracture
8. Serious active infection requiring IV antibiotics and/or hospitalization within 7 days of enrollment
9. Known severe hypersensitivity to any of the study drugs or excipients, including history of allergic, anaphylactic, or other severe hypersensitivity reactions to fusion proteins, products containing Cremophor EL (eg, cyclosporin for injection concentrate and teniposide for injection concentrate)
10. Require regular blood transfusions, platelet transfusions, or granulocyte colony stimulating factor.
11. For female patients of childbearing potential, the following are exclusion criteria, as applicable:
12. Refusal to use highly effective method of contraception or to practice true abstinence during treatment and for 6 months after the last dose of study drug
13. Pregnant or breast feeding;
14. Presence of any other condition that may increase the risk associated with enrollment on the study, interfere with data interpretation, or make the patient inappropriate for study enrollment in the opinion of the treating investigator
15. Prior treatment with or participation in a study with BMX-001
16. A history of additional risk factors for Torsades de Pointes (e.g., congestive heart failure, hypokalemia, known family history of Long QT Syndrome).
17. Severe, active co-morbidity, as defined in protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
To determine the Recommended Phase 2 Dose of BMX-001 in combination with paclitaxel in a safety cohort of patients. This would be carried forward as the dose to be used in the expanded cohort portion of the trial. | 8 weeks
  The metric used to characterize the primary outcome measure is the determination of the Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) of BMX-001 when administered in combination with paclitaxel. This will be based on the incidence of Dose- Limiting Toxicities (DLTs) observed in a safety cohort (dose escalation design) of patients over an 8-week period. The RP2D will be identified as the highest dose level at which a predefined acceptable DLT rate is observed, and this dose will be carried forward for use in the expanded cohort portion of the trial. We seek to determine if the current dose used in previous clinical trials dose can be safely doubled by giving two 28 mg doses s.c. that are 4-6 hours apart given on the first day of each week to optimize the opportunity for achieving efficacy.

SECONDARY OUTCOMES:
To evaluate preliminary efficacy based on objective response rate (ORR) using RECIST v 1.1 per investigator assessment on all evaluable subjects enrolled | 1 year
  The metric used to characterize the secondary outcome measure is the Objective Response Rate (ORR), which will be assessed using RECIST v1.1 criteria. This will be measured as the proportion of evaluable subjects who achieve a complete or partial response to the treatment as determined by the investigator. Evaluations will be conducted at baseline, post-treatment at every 8- week interval during the first 48 weeks following treatment initiation (Cycle 1, Day 1), and every 12 weeks thereafter until disease progression or study termination.
To evaluate preliminary efficacy based on progression free survival (PFS) using RECIST v 1.1 per investigator assessment on all evaluable subjects enrolled | 1 year
  The metric used to characterize the secondary outcome measure is the Progression Free Survival (PFS) which will be assessed using RECIST v1.1 criteria. This will be measured as the proportion of evaluable subjects who achieve a complete or partial response to the treatment as determined by the investigator. Evaluations will be conducted at baseline, post-treatment at every 8- week interval during the first 48 weeks following treatment initiation (Cycle 1, Day 1), and every 12 weeks thereafter until disease progression or study termination.
To describe patient-reported outcomes of health related quality of life (HRQoL) using Functional Assessment of Cancer Therapy/Gynecologic Oncology - Neurotoxicity (FACT/GOG-NTX) Questionnaire and monofilament testing | 1 year
  The metric used to characterize this secondary outcome measure is patient-reported outcomes (PRO) related to health-related quality of life (HRQoL) and overall quality of life (QoL). These outcomes will be assessed using the FACT/GOGNTX Questionnaire and monofilament testing.
  Measurements will be taken at baseline and then every 28 days until disease progression. The assessments will provide insights into the impact of the treatment on patients' physical, emotional, and functional well-being, as well as the extent of peripheral neuropathy experienced during the study.

OTHER OUTCOMES:
To characterize the Cmax of BMX-001 when delivered in combination with PTX in recurrent ovarian or endometrial cancer in all evaluable subjects enrolled. | 2 weeks
  The metric used to characterize this outcome measure is Cmax of BMX-001 when administered in combination with paclitaxel (PTX) in patients with recurrent ovarian or endometrial cancer.
  Pharmcaokinetic samples will be collected on Day 1 and Day 8 at pre-dose, and at 30 minutes, 1 hour, and 2 hours postdose. For Dose Levels 2 and 3 (with two doses of BMX-001 per day), samples will be collected on Day 1 and Day 8 at pre-dose, 30 minutes, 1 hour, and 4-6 hours post-dose, and then at 30 minutes and 1 hour post-second dose.
To characterize the Tmax and half life of BMX-001 when delivered in combination with PTX in recurrent ovarian or endometrial cancer in all evaluable subjects enrolled. | 2 weeks
  The metric used to characterize this outcome measure is Tmax and half-life of BMX-001 when administered in combination with paclitaxel (PTX) in patients with recurrent ovarian or endometrial cancer.
  Pharmacokinetic samples will be collected on Day 1 and Day 8 at pre-dose, and at 30 minutes, 1 hour, and 2 hours postdose. For Dose Levels 2 and 3 (with two doses of BMX-001 per day), samples will be collected on Day 1 and Day 8 at pre-dose, 30 minutes, 1 hour, and 4-6 hours post-dose, and then at 30 minutes and 1 hour post-second dose.
To characterize the area under the plasma concentration versus time curve of BMX-001 when delivered in combination with PTX in recurrent ovarian or endometrial cancer in all evaluable subjects enrolled. | 2 weeks
  The metric used to characterize this outcome measure is the area under the plasma concentration versus time curve (AUC) of BMX-001 when administered in combination with paclitaxel (PTX) in patients with recurrent ovarian or endometrial cancer.
  Pharmacokinetics samples will be collected on Day 1 and Day 8 at pre-dose, and at 30 minutes, 1 hour, and 2 hours postdose. For Dose Levels 2 and 3 (with two doses of BMX-001 per day), samples will be collected on Day 1 and Day 8 at pre-dose, 30 minutes, 1 hour, and 4-6 hours post-dose, and then at 30 minutes and 1 hour post-second dose.
To assess correlations between B cell lymphoma/ leukemia 2 (BCL2), Nrf2, TNF- # and NFkB RNA and protein expression and activation, ctDNA, and clinical endpoints (response and progressionfree survival) in all evaluable subjects enrolled | 1 year
  The metric used to characterize this outcome measure is the correlation between molecular biomarkers and clinical outcomes. Specifically, the study will assess the expression and activation levels of B cell lymphoma/leukemia 2 (BCL2), Nrf2, TNF-alpha, and NFkB RNA and proteins, as well as circulating tumor DNA (ctDNA). These molecular data will be correlated with clinical endpoints, including response to treatment (ORR) and progression-free survival (PFS). Samples will be collected at baseline and post-treatment to evaluate these associations in all evaluable subjects. This analysis aims to identify potential biomarkers that could predict treatment efficacy and disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: James Crapo, MD, Study Director — BioMimetix JV, LLC; Angeles Secord, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided